CLINICAL TRIAL: NCT04528004
Title: Mechanistic Studies of Nicotinamide Riboside in Human Heart Failure
Acronym: NRII
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kevin O'Brien, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00007432; 1R01HL144937-01A1 (NIH)
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure, Systolic; Heart Failure NYHA Class IV; Metabolic Disturbance
MeSH Terms: conditions — Heart Failure, Systolic | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized, interventional trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization with a 2:1 nicotinamide riboside:matching placebo allocation ratio. Dispensing of nicotinamide riboside and matching placebo will be performed by the University of Washington Investigational Drug Services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotinamide riboside (Experimental): Participants randomized to Nicotinamide Riboside (NR) and scheduled to receive an LVAD will receive nicotinamide riboside (NR) capsules according to the following administration schedule:
  Dose Escalation Day 1: 250 mg (1 capsule) twice daily (total daily intake = 500 mg) Day 2: 500 mg (2 capsules) twice daily (total daily intake = 1000 mg) Day 3: 1000 mg (4 capsules) twice daily (total daily intake = 2000 mg) Dose Maintenance Day 4: 1000 mg (4 capsules) twice daily Day 5-14 as applicable thru Day Before Surgery: 1000 mg (4 capsules) twice daily Washout Day of LVAD Surgery and/or Day 15: None
  Interventions: Drug: Nicotinamide riboside
- Placebo (Placebo Comparator): Participants randomized to Placebo and scheduled to receive an LVAD will receive Placebo capsules according to the following administration schedule:
  Dose Escalation Day 1: 250 mg (1 capsule) twice daily (total daily intake = 500 mg) Day 2: 500 mg (2 capsules) twice daily (total daily intake = 1000 mg) Day 3: 1000 mg (4 capsules) twice daily (total daily intake = 2000 mg) Dose Maintenance Day 4: 1000 mg (4 capsules) twice daily Day 5-14 as applicable thru Day Before Surgery: 1000 mg (4 capsules) twice daily Washout Day of LVAD Surgery and/or Day 15: None
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotinamide riboside — Nicotinamide riboside 250mg capsules
  Arms: Nicotinamide riboside
Other: Placebo — Matching placebo 250mg capsules
  Arms: Placebo

SUMMARY:
Preliminary animal studies by ourselves and others suggest that the dietary supplement, nicotinamide riboside (NR), may improve cardiac function in heart failure (HF) by increasing cellular levels of its metabolite, nicotinamide adenine dinucleotide (NAD+, NADH). This Study will address a key gap in current knowledge by assessing the mechanisms through which raising blood and myocardial NAD+ levels in humans mediates changes in mitochondrial function, protein and epigenetic modifications, as well as inflammation. Human myocardium will be obtained after 4-14 days of oral NR supplementation from advanced heart failure patients undergoing elective left ventricular assist device (LVAD) implantation. Positive results would provide evidence to proceed with further studies of NR as a mitochondria-targeted metabolic therapy in heart failure.

DETAILED DESCRIPTION:
To definitively demonstrate the effects of increasing NAD+ levels in HF patients, this randomized, placebo-controlled trial of NR in 40 participants scheduled for elective LVAD surgery with the underlying hypotheses that those randomized to NR will have higher myocardial NAD+ levels, improved mitochondrial function, restored gene expression and reduced inflammatory response as compared to participants randomized to placebo. To this end, the study has the following specific aims:

Aim 1: Randomize 40 participants undergoing elective LVAD placement into a double-blind, placebo-controlled study of NR vs. placebo at an NR:placebo ratio of 2:1.

1. Participants will have labs (including safety panels) drawn at baseline (Day 1), with NR or placebo dose escalation to 1000mg twice daily by Day 3, and the last dose administered the evening prior to surgery.
2. Final labs will be drawn on the day of surgery, and samples of fresh cardiac tissue removed from the left ventricular apex during LVAD implantation surgery will be collected in the operating room.

Aim 2: Determine the effect of NR vs. placebo on NAD(H) levels, mitochondrial function and its regulation through epigenetic modifications in the failing myocardium.

1. Measure NAD+ and NADH levels in the blood and myocardium of the participants.
2. Assess mitochondrial morphology and function in cardiac tissue using electron microscopy (EM) and isolated mitochondria.
3. Determine changes in protein acetylation in the mitochondrial and non-mitochondrial compartments and in nuclear gene regulation.

Aim 3: Test the hypothesis that NR improves mitochondrial function and reduces inflammatory response in HF patients.

1. Measure mitochondrial function in peripheral blood mononucleated cells (PBMC).
2. Determine the inflammatory response in PBMC from NR-treated vs. placebo participants.
3. Compare effects on the circulating inflammasome vs. myocardial inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. End-stage heart failure due to ischemic or non-ischemic cardiomyopathy

   a. If implanted for destination therapy indication, must have New Your Heart Association (NYHA) Class IV Heart Failure AND left ventricular ejection fraction (LVEF) <25% OR maximum minute consumption of oxygen (VO2) <14 OR on requirement for continuous intravenous inotropes
2. Meet clinical and socioeconomic screening criteria for elective LVAD implantation by the University of Washington Mechanical Circulatory Support Program
3. Scheduled (or soon to be scheduled) for elective LVAD implantation
4. Age >18 years

Exclusion Criteria:

1. End-stage heart failure due to causes other than ischemic or non-ischemic cardiomyopathy (e.g., valvular, hypertrophic or infiltrative cardiomyopathies).
2. Disease that disqualifies from consideration for LVAD implantation by the University of Washington program:

   1. Cirrhosis as evidenced by liver biopsy
   2. Irreversible, severe renal disease (estimated glomerular filtration rate (eGFR) <30) or on chronic dialysis
   3. Untreated thyroid disease (hyper- or hypo-thyroidism)
   4. Severe complications of diabetes, such as diabetes-related amputation, severe retinopathy, peripheral neuropathy or diabetic renal disease (eGFR <30)
3. Tissue physiology or other factors that, in the opinion of the Cardiac Surgeons, make the patient at unacceptably high risk for adverse outcomes.
4. Non-compliance with current treatments, including failure to follow prescribed therapies, such as medications, clinic visits, diagnostic testing and behavioral contracts
5. Active use/abuse of illicit substances
6. Lack of adequate caregiver support to help patient manage LVAD
7. Known allergies to niacin, nicotinamide or warfarin
8. Inability to perform Study visits or procedures
9. Unwillingness/inability to provide informed consent.
10. Participants considered by the attending cardiologist and/or the investigator to be unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-26 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Between-group comparisons of whole blood NAD+ levels | Up to 14 days
  Comparisons of whole blood NAD+ levels on the Day of LVAD Surgery in participants randomized to NR vs. placebo

SECONDARY OUTCOMES:
Between-group comparisons of myocardial NAD(H) levels | Up to 14 days
  Comparisons of myocardial NAD(H) levels in participants randomized to NR vs. placebo
Between-group comparisons of myocardial mitochondrial respiratory function. | Up to 14 days
  Comparisons of myocardial mitochondrial respiration in participants randomized to NR vs. placebo
Between-group comparisons of myocardial mitochondrial morphology. | Up to 14 days
  Comparisons of myocardial mitochondrial morphology, by electron microscopy, in participants randomized to NR vs. placebo
Between-group comparisons of myocardial protein acetylation | Up to 14 days
  Comparisons of myocardial protein acetylation in participants randomized to NR vs. placebo
Between-group comparisons of myocardial gene expression by RNA-seq and the myocardial epigenome by ATAC-seq | Up to 14 days
  Comparisons, NR vs. placebo-treated participants, of myocardial gene expression by RNA sequencing (RNA-seq) and the myocardial epigenome by the Assay for Transposase-Accessible Chromatin using sequencing (ATAC-seq)
Between-group comparisons of inflammatory markers in blood | Up to 14 days
  Comparisons, in patients randomized to NR vs. placebo of: 1) plasma levels of highly-sensitive C-reactive protein, interleukin-1beta, interleukin-6, interleukin-18, tumor necrosis factor-alpha, and NLR family pyrin domain containing 3 (NLRP3), as well as 2) mRNA expression of these cytokines in isolated peripheral blood mononuclear cells
Between-group comparisons of inflammatory markers in myocardium | Up to 14 days
  Comparisons by quantitative morphometry of immunohistochemical staining of macrophages (including M1 and M2 phenotypes) in myocardium in participants randomized to NR vs. placebo

OTHER OUTCOMES:
Correlations of whole blood NAD+ levels with secondary outcome measures | Up to 14 days
  Analyses of correlations of whole blood NAD+ levels and their changes with each of the secondary outcome measures in the NR-treated group
Correlations of myocardial NAD(H) levels with secondary outcome measures | Up to 14 days
  Analyses of correlations of myocardial NAD(H) levels and their changes with secondary outcome measures in the NR-treated group

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D O'Brien, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The Investigators plan to deposit study results in BioLINCC. The Study will generate data that is primarily applicable to the basic research questions that are proposed. It is the explicit intention of the Investigators that these data will be placed in a readily accessible public database. The Investigators anticipate placing de-identified study results into the NHLBI data repository at the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) (biolincc.nhlbi.nih.gov/home/). Data sets will be submitted no later than three years after the final study dataset is locked or two years after the core manuscript from the trial has been published, whichever comes first.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be deposited no later than three years after the final study dataset is locked or two years after the core manuscript from the trial has been published, whichever comes first.
Access Criteria: It is the explicit intention of the Investigators that these data will be placed in a readily accessible public database. The Investigators anticipate placing de-identified study results into the NHLBI data repository at the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) (biolincc.nhlbi.nih.gov/home/).

DOCUMENTS (1):
  • Informed Consent Form (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT04528004/ICF_000.pdf